CLINICAL TRIAL: NCT02056717
Title: The Effect of Dexamethasone on Inflammatory Response After Uterine Artery Embolization
Brief Title: Use of Dexamethasone in Uterine Artery Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2013-0863
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Uterine Myoma; Adenomyosis
MeSH Terms: conditions — Myofibroma; Adenomyosis | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone group (Experimental)
  Interventions: Drug: Dexamethasone
- Control group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Administration of dexamethasone 10 mg IV 1 h before UAE
  Arms: Dexamethasone group
Drug: Normal saline — Administration of normal saline 2 mL IV 1 h before UAE
  Arms: Control group

SUMMARY:
The primary purpose of this study is to investigate the effects of dexamethasone on inflammatory reactions after uterine artery embolization. The secondary purpose of this study it to investigate the effects of dexamethasone on postembolization syndrome (severe pain, nasea and vomiting).

ELIGIBILITY:
Inclusion Criteria:

* Uterine artery embolization due to multiple myoma or adenomyosis

Exclusion Criteria:

* Diabetic mellitus
* Steroid administration
* Liver or kidney dysfuntion
* High baseline CRP or leukocytosis (>11,000/μL )
* Drug allergy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Inflammatory reactions | 24 hours
  CRP, WBC, neutrophil (%), cortisol : pre-UAE, post-UAE 12 h, post-UAE-24 h IL-6 : pre-UAE, post-UAE-24 h

SECONDARY OUTCOMES:
Pain | 24 hours
  Immediately after UAE, post-UAE 1, 2, 4, 6, 8, 12, 24 h
Nausea and vomiting | 24 hours
  Immediately after UAE, post-UAE 1, 2, 4, 6, 8, 12, 24 h
Sucessful rate at 3 month after UAE | 3 month
  Utrerine volume and complete necrosis incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea